CLINICAL TRIAL: NCT03131726
Title: Treatment of Graves´ophthalmopathy with Simvastatin (GO-S)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tereza Planck
Record Dates: First submitted 2017-03-10; First posted 2017-04-27 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Graves Ophthalmopathy; Thyroid Associated Ophthalmopathy; Thyroid Associated Orbitopathy
Keywords: simvastatin; diclofenac
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Experimental): simvastatin 40 mg daily for 6 months
  Interventions: Drug: Simvastatin 40mg
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: Simvastatin 40mg — see arm description
  Other Names: ATC-code: C10AA01
  Arms: Simvastatin

SUMMARY:
In an investigator initiated multicenter trial (Malmö, Odense, Århus) the investigators aim at evaluating activity of Graves´ophthalmopathy (GO) and progress to severe GO in patients with mild to moderate Graves´ ophthalmopathy treated with simvastatin or no treatment.

DETAILED DESCRIPTION:
Progression of GO from mild-moderate to severe disease:

Criteria for start of treatment with corticosteroids, retrobulbar irradiation, or orbital decompression are severe soft tissue swelling (NO SPECS class 2c), risk of corneal ulcers with or without exophthalmos, double vision within 30 degrees, and optic nerve dysfunction. Patients who progress will be followed until the end of the study with the ongoing randomized treatment.

Withdrawal criteria:

1. Patients may withdraw from the trial at any time without any consequences for their future treatment.
2. Patients may be withdrawn from the trial at the discretion of the investigator if judged to be non-compliant with trial procedures or due to safety concerns.
3. Patients must be withdrawn from the trial if they become pregnant or develop congestive heart failure, renal insufficiency, coagulopathy, gastric ulcer, inflammatory bowel disease, diabetic retinopathy, diabetic nephropathy, severe myopathy, or rhabdomyolysis.

Laboratory investigations before randomization:

TSH, fT4, fT3, TRAb, TPOAb, p-glucose, HbA1c, creatinine or cystatin C for estimation of GFR according to the routines of the individual study centers. Biobank samples for analysis of potential markers of ophthalmopathy, DNA (buffy coat), RNA (whole blood), serum, and plasma according to separate sampling instructions.

Clinical appointments and treatment of ophthalmopathy:

Endocrinologist and ophthalmologist judge the presence of ophthalmopathy in patients with Graves´ disease and asses inclusion and exclusion criteria before randomization to treatment with or without simvastatin.

The activity of ophthalmopathy is judged according to CAS (clinical activity score) and registered by the ophthalmologist:

Spontaneous retrobulbar pain 0. No 1. Yes Painful eye-movements 0. No 1, Yes Eye lid erythema 0. No 1. Yes Conjunctival injection 0. No 1. Yes Chemosis 0. No 1. Yes Swollen caruncula 0. No 1. Yes Eye lid edema or swelling 0. No 1, Yes Sum (points)

In parallel, evaluation with modified CAS is performed and registered by the ophthalmologist:

Spontaneous retrobulbar pain 0. No 1. Mild 2. Moderate 3. Severe Painful eye-movements 0. No 1. Mild 2. Moderate 3. Severe Eye lid erythema 0. No 1. Mild 2. Moderate 3. Severe Conjunctival injection 0. No 1. Mild 2. Moderate 3. Severe Chemosis 0. No 1. Mild 2. Moderate 3. Severe Swollen caruncula 0. No 1. Mild 2. Moderate 3. Severe Eye lid edema or swelling 0. No 1. Mild 2. Moderate 3. Severe Sum (points)

Severity is judged by the following parameters and registered in the ophthalmologist´s protocol: vision, sense of colour, eye papillae edema, eye protrusion, impaired eye movements, corneal ulcers.

Judgement of thyroid function and ophthalmopathy is performed by an endocrinologist/ophthalmologist at inclusion and after 3 and 6 months. The ophthalmologist who evaluates activity and severity of ophthalmopathy is not aware of which treatment arm (simvastatin or control) the patient has been randomized to (single-blind design).

Patients are photographed at each visit and every fifth photograph of ophthalmopathy status is sent to the other centers for evaluation of selected parameters in CAS to evaluate the inter-observer variation.

All patients who fulfill the inclusion criteria and lack exclusion criteria and have signed informed consent will be randomized to treatment simvastatin 40 mg 1x1 or no additional treatment for 6 months. Drugs for treatment are prescribed for 3 months and repeated at control visits. Information on collection of drugs is checked with lists obtained from the pharmacy.

Thyroid treatment:

Patients with Graves ´ hyperthyroidism are treated with ATD. This can be done with the block and replace approach or by titration of ATD according to the local tradition as long as euthyroidism is achieved during the study period (normal fT4 and fT3 with TSH below the upper limit of the local reference interval).

Patients with clinical ophthalmopathy at diagnosis can be included no earlier than 2 months after treatment with ATD and only if biochemical or clinical euthyroidism has been achieved.

Patients who have stopped medication with ATD can be included at the earliest after 2 months and only if clinically and biochemically euthyroid.

Patients who have been treated with radioiodine can be included 6 months after radioiodine if euthyroid. In case of hypothyroidism, patients must be treated with L-thyroxine and be clinically and biochemically euthyroid before inclusion.

Patients who have had thyroidectomy can be included when euthyroidism has been achieved with L-thyroxine.

Statistical considerations and study design:

The primary evaluation variable is change in CAS after 6 months. If it is assumed that the spontaneous change without treatment is -0.6 and if the treatment groups improvement in CAS is -1.9, 34 patients in each group are needed to achieve 80 % power at significance level of 0.05. The basis of this calculation is a study on the effects of selenium treatment in patients with mild to moderate ophthalmopathy (Marcocci 2011).

The investigators will stratify for smoking at randomization which will be performed in blocks of 6 within each participating center.

The secondary exclusion and lost to follow-up rate of patients is estimated to 10 % during the study period. The investigators therefore plan to include a total of 80 patients. The following reasons are expected to cause secondary exclusion/ loss of patients:

1. Side effects of treatment
2. Lack of compliance or safety routines not being followed

Ethics:

All patients will receive written information on treatment alternatives, possible side-effects of any drugs used, and the aim of the study which has been approved by relevant ethics committees.

Publication and authorship:

The primary results will be reported in an appropriate medical journal after discussion with the participants of the study and authorship can be claimed if the participant has included at least 10 % of the total number of patients.

Visit schedule:

S = Screening tests, TSH, fT4, fT3, TRAb, TPOAb, Hb, fasting- p-glucose, HbA1c, eGFR (creatinine and cystatin C), ASAT, ALAT, ALP, GT, CK, cholesterol, triglycerides R = Routine tests, TSH, fT4, fT3, Hb, eGFR, CK, ASAT, ALAT, ALP, GT, cholesterol, triglycerides, TRAb, anti-TPO B = Biobank samples according to separate instructions C = Clinical control - vital signs, physical examination, eye status O = Ophthalmologist - eye status, OCT of conjunctive Q = Quality of life questionnaire (SF36,ThyrPro and GO-QoL)

Time 0 S, B, C, O, Q 3 months S, B, C, O, Q 6 months S, B, C, O, Q

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Active mild to moderate with at least one sign of mild GO (NO SPECS class 2a and b) with reference to Colour Atlas at EUGOGO website (www.eugogo.eu). Exophthalmos up to 24 mm with a disease duration of <18 months (as recorded by the patient)
3. Graves´ disease with clinical and laboratory euthyroidism after stopping treatment with anti thyroid drugs (ATD), or 2 months treatment with ATD, or euthyroid 6 months after treatment with radioiodine, or euthyroid after total thyroidectomy. Clinical and laboratory euthyroidism is defined as normal fT4, fT3 and TSH below the upper limit of the local reference interval and no clinical symptoms or signs of hyperthyroidism. L-thyroxine is used to achieve euthyroidism during the study period.

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Previous treatment of Graves´ ophthalmopathy
3. Severe Graves ophthalmopathy requiring corticosteroid treatment, retrobulbar irradiation, orbital decompression surgery
4. Current or previous treatment with simvastatin or other statins (within 3 months)
5. Allergy (skin rash or systemic reactions) to statins
6. Congestive heart failure
7. Renal insufficiency (glomerular filtration rate <60 ml/min)
8. ASAT or ALAT > 2.5 times the upper limit of the local laboratory
9. Alcoholism as judged by local criteria
10. Coagulopathy including treatment with warfarin or new oral anti-coagulation drugs
11. Previous or current gastric ulcer
12. Inflammatory bowel disease diabetic retinopathy or nephropathy
13. Trauma within 10 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical activity score (CAS) after 6 months | 6 months
  Change in 7-point clinical activity score (CAS) after 6 months treatment with simvastatin or no treatment
Number of patients with progression to severe GO during 6 months | 6 months
  Number of patients with progression to severe GO in each group (simvastatin, no treatment) during 6 months treatment

SECONDARY OUTCOMES:
Change in Modified Clinical activity score | 3 and 6 months
  Change in Modified clinical activity score after 3 and 6 months treatment with simvastatin or no treatment
Optical coherence tomography | 3 and 6 months
  Evaluation of conjunctival thickness with optical coherence tomography after 3 and 6 months treatment with simvastatin or no treatment
Quality of life with SF36 | 6 months
  Quality of life after 6 months treatment with simvastatin or no treatment assessed with the SF36 questionnaire
Quality of life with ThyrPro | 6 months
  Quality of life after 6 months treatment with simvastatin or no treatment assessed with the ThyPro questionnaire
Quality of life with GO-QoL | 6 months
  Quality of life after 6 months treatment with simvastatin or no treatment assessed with the GO-QoL questionnaire
TRAb | 3 and 6 months
  TRAb after 3 and 6 months treatment with simvastatin or no treatment
TPO-Ab | 3 and 6 months
  TPOAb after 3 and 6 months treatment with simvastatin or no treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Planck, MD, PhD, Principal Investigator — Lund University and Skåne University Hospital
Locations (1):
- Dpt. of Endocrinology, SUS Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided